CLINICAL TRIAL: NCT07261670
Title: A Comparative Study of Virtual Reality and Sensory-Adapted Dental Environments for Dental Anxiety Reduction in Individuals With Borderline Intellectual Functioning
Brief Title: A Comparative Study of Virtual Reality and Sensory-Adapted Dental Environments for Dental Anxiety Reduction in Individuals With BIF
Acronym: VR-SADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oasi Research Institute-IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-2794677_
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Borderline Intellectual Functioning (BIF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): immersive VR software delivered through Meta Quest 3® headset during dental procedure
  Interventions: Device: Virtual Reality Distraction - immersive VR software delivered through Meta Quest 3® headset during dental procedure
- Sensory adapted dentist environment Control (Active Comparator): Sensory adapted dentist environment designed to reduce sensory stimuli with:
  * soft and dim lighting
  * a screen projecting familiar movies, cartoons, or videos previously provided by the family
  * a dental turbine handpiece covered with a sponge layer to minimize noise
  Interventions: Device: Sensory adapted dentist environment

INTERVENTIONS:
Device: Virtual Reality Distraction - immersive VR software delivered through Meta Quest 3® headset during dental procedure — immersive VR software delivered through Meta Quest 3® headset during dental procedure
  Arms: Virtual Reality Distraction
Device: Sensory adapted dentist environment — Sensory adapted dentist environment designed to reduce sensory stimuli with: - soft and dim lighting - a screen projecting familiar movies, cartoons, or videos previously provided by the family - a dental turbine handpiece covered with a sponge layer to minimize noise
  Arms: Sensory adapted dentist environment Control

SUMMARY:
A randomized clinical trial was conducted with 98 participants with borderline intellectual functioning (BIF) and moderate dental anxiety (DAS: 9-12). Participants were assigned in a 1:1 ratio to either the Virtual reality (VR) or sensory adapted dentist environment (SADE) group (49 per group). The primary outcome was treatment success, defined as completing a dental restoration under local anesthesia within 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age of participants between 10 and 13 years
* Diagnosis of Borderline Intellectual Func-tioning (BIF) confirmed by experienced neuropsychiatrists according to DSM-5 criteria
* Moderate dental anxiety, defined by a DAS score between 9 and 12
* Presence of at least one tooth with a Class I carious lesion requiring restorative treatment

Exclusion Criteria:

* absence of dental anxiety (DAS score = 4)
* the presence of mild anxiety (DAS score = 5-8)
* high or severe anxiety (DAS score ≥ 13)

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment success | Duration of procedure
  Completion of restorative dental procedure under local anesthesia within 30 minutes and positive overall treatment experience (dichotomous: success vs. failure)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ass. Oasi Maria SS, Troina, EN, Italy

IPD SHARING:
Plan to Share IPD: Undecided